CLINICAL TRIAL: NCT06311981
Title: A Prospective Phase II Clinical Study of Carbon Ion Radiotherapy for Locally Advanced Non-small Cell Lung Cancer in the Older Adult
Brief Title: Carbon Ion Radiotherapy for Locally Advanced Lung Cancer in Elderly Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jian Chen (Other)
Responsible Party: Sponsor-Investigator, Jian Chen, Clinical Professor, Shanghai Proton and Heavy Ion Center
Organization: Shanghai Proton and Heavy Ion Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPHIC-TR-THLC2023-08
Record Dates: First submitted 2024-03-09; First posted 2024-03-15 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Non-small Cell Lung Cancer; Older People; Carbon Ion Radiotherapy; Radiotherapy Side Effect
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Radiation Injuries | interventions — Heavy Ion Radiotherapy; Base Sequence; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study arm (Experimental): The patient will receive carbon ion radiotherapy with 70Gy per 20 fractions. Patients with genetic mutations (including but not limited to EGFR, ALK, etc.) should receive targeted therapy as their systemic therapy. For patients who are not suitable for targeted therapy, we recommend single regimen chemotherapy in sequence with radiotherapy. The drugs include etoposide, platinum (carboplatin, cisplatin, nedaplatin or loplatin), vinorelbine, paclitaxel (including liposome paclitaxel and albumin paclitaxel), docetaxel, pemetrexel, gemcitabine, etc. If there is no contraindication to PD-1/PD-L1 immunotherapy, it can be combined with immunotherapy, such as Pembrolizumab. For patients who cannot tolerate chemotherapy, PD-1/PD-L1 immunotherapy is recommended. The progression-free survival rate, toxicity, local control rate, cause-specific survival rate and overall survival rate were observed with regular follow-up after treatment.
  Interventions: Radiation: carbon ion radiotherapy; Other: targeted therapy; Other: single regimen chemotherapy in sequence with radiotherapy

INTERVENTIONS:
Radiation: carbon ion radiotherapy — The patient will receive carbon ion radiotherapy with 70Gy per 20 fractions. Patients with genetic mutations (including but not limited to EGFR, ALK, etc.) should receive targeted therapy as their systemic therapy. For patients who are not suitable for targeted therapy, we recommend single regimen chemotherapy in sequence with radiotherapy. The drugs include etoposide, platinum (carboplatin, cisplatin, nedaplatin or loplatin), vinorelbine, paclitaxel (including liposome paclitaxel and albumin paclitaxel), docetaxel, pemetrexel, gemcitabine, etc. If there is no contraindication to PD-1/PD-L1 immunotherapy, it can be combined with immunotherapy, such as Pembrolizumab. For patients who cannot tolerate chemotherapy, PD-1/PD-L1 immunotherapy is recommended. The progression-free survival rate, toxicity, local control rate, cause-specific survival rate and overall survival rate were observed with regular follow-up after treatment.
Other: targeted therapy — targeted therapy
Other: single regimen chemotherapy in sequence with radiotherapy — single regimen chemotherapy in sequence with radiotherapy

SUMMARY:
To observe the effect and toxicity of carbon ion radiotherapy on local advanced non-small cell lung cancer over 75 years old patients. Systemic therapy could be targeted therapy, chemotherapy or immunotherapy.

DETAILED DESCRIPTION:
The patient will receive carbon ion radiotherapy with 70Gy per 20 fractions. Patients with genetic mutations (including but not limited to EGFR, ALK, etc.) should receive targeted therapy as their systemic therapy. For patients who are not suitable for targeted therapy, we recommend single regimen chemotherapy in sequence with radiotherapy. The drugs include etoposide, platinum (carboplatin, cisplatin, nedaplatin or loplatin), vinorelbine, paclitaxel (including liposome paclitaxel and albumin paclitaxel), docetaxel, pemetrexel, gemcitabine, etc. If there is no contraindication to PD-1/PD-L1 immunotherapy, it can be combined with immunotherapy, such as Pembrolizumab. For patients who cannot tolerate chemotherapy, PD-1/PD-L1 immunotherapy is recommended. The progression-free survival rate, toxicity, local control rate, cause-specific survival rate and overall survival rate were observed with regular follow-up after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Older than 75 years old.
* ECOG general status score of 0-2.
* Primary non-small cell lung cancer (NSCLC) confirmed by histology or cytological pathology, T1-4N1-3M0, stage IIb-IIIc (AJCC/UICC 8th edition).
* Medically inoperable, or patient refuses surgery.
* Adequate organ function: 1). Blood function: absolute neutrophil count (ANC) ≥1.5 x 109/L, platelet count ≥80 x 109/L, hemoglobin ≥9 g/dL 2). Lung function: FEV1>25%, DLCO>25% 3). Cardiac function: no serious pulmonary hypertension, cardiovascular and cerebrovascular diseases, peripheral vascular diseases, serious chronic heart disease and other complications that may affect radiotherapy.4). Adequate liver function: total bilirubin <1.5 times the upper limit of normal value, and AST, ALT<2 times the upper limit of normal value. 5). Adequate renal function: serum creatinine ≤1.5 times the upper limit of normal or calculated creatinine clearance ≥50 ml /min, and urinary protein <2+. Patients with a baseline urinary protein level of 2+ or more should have a 24-hour urine collection and evidence of a 24-hour urinary protein level of 1g or less.
* Sign informed consent.

Exclusion Criteria:

* Patient with squamous cell carcinoma was treated with bevacizumab before carbon ion radiotherapy.
* Complicated with other malignant tumors that have not been controlled.
* Patient whose particle radiotherapy plan cannot meet the minimum target dose coverage and dose volume limitation requirements, or cannot meet the dose constrains of normal tissue or organs.
* Chest radiation therapy or radioactive particle implantation history.
* Cardiac pacemakers or other internal metal prosthesis implants that may be affected by high-energy radiation or may affect the dose distribution to the radiation target area.
* HIV positive. Hepatitis virus replication phase, need to receive antiviral therapy, but because of concomitant disease cannot receive antiviral therapy. Active stage of syphilis.
* A history of mental illness may hinder the completion of treatment.
* With serious comorbidity that may interfere with radiotherapy, including: (a) Acute infectious diseases or acute active phase of chronic infection. b) Unstable angina pectoris, congestive heart failure, myocardial infarction that has been hospitalized in the past 6 months. c) Exacerbations of chronic obstructive pulmonary disease or other respiratory conditions requiring hospitalization. d) Severely impaired immune function. e) Diseases with excessive sensitivity to radiation such as ataxia telangiectasia. f) Other diseases that may affect particle radiotherapy.
* Other circumstances that the physician considers inappropriate to participate in clinical study.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2025-06-17 (Estimated); Study Completion 2026-06-17 (Estimated)

PRIMARY OUTCOMES:
Disease progression-free survival rate | From date of radiotherapy started until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.
  Disease progression-free survival rate was defined from the start of carbon ion radiotherapy till the date of disease progression at any site or death, or the last follow up.
Incidence of Treatment-induced Adverse Events | From date of radiotherapy started, every 3-4 months within the first 2 years, every 6 months between years 3 and 5, and annually thereafter, assessed up to 100 months.
  Treatment-induced toxicities were scored using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, for events observed after the first dose of irradiation. Toxicities occurred 90 or more days after the completion of CIRT were defined as late toxicities.

SECONDARY OUTCOMES:
Local control rate | From date of radiotherapy started until the date of first documented local disease progression, assessed up to 100 months.
  Local control rate was defined from the start of carbon ion radiotherapy till the date of local failure or the last follow-up
Cause-specific survival rate | From date of radiotherapy started until the date of first documented death caused by non-small cell lung cancer treated in this study, assessed up to 100 months.
  Cause-specific survival rate was defined from the start of carbon ion radiotherapy till the date of death caused by non-small cell lung cancer treated in this study or the last follow-up
Overall survival rate | From date of radiotherapy started until the date of death from any cause, assessed up to 100 months.
  Overall survival rate was defined from the start of carbon ion radiotherapy till the date of death or the last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Jingfang Mao, PHD, Principal Investigator — Shanghai Proton and Heavy Ion Center
Locations (1):
- Shanghai Proton and Heavy Ion Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided